CLINICAL TRIAL: NCT02485795
Title: A Multicenter Longitudinal Observational Study Evaluating Genotypic Association wIth Clinical Outcomes in Interventional Pain Management Modalities
Brief Title: Observational Study of the Impact of Genetic Testing on Healthcare Decisions and Care in Interventional Pain Management
Acronym: MOSAIC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Proove Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PB007
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Pain; Chronic Pain; Back Pain; Nociceptive Pain; Neuropathic Pain; Musculoskeletal Pain; Neck Pain; Pain, Intractable
Keywords: Pain Management; Genetic Variation; Genetic Polymorphism; Polymorphism, Single Nucleotide Genetic Association Studies; Healthcare Utilization
MeSH Terms: conditions — Pain; Chronic Pain; Back Pain; Nociceptive Pain; Neuralgia; Musculoskeletal Pain; Neck Pain; Pain, Intractable; Agnosia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pain patients: Observational; Patients presenting to interventional pain management centers for therapy.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — This study will evaluate the impact of genetic testing information on medical regimen plans and whether this information results in benefits to patient care.

SUMMARY:
The purpose of this study is to evaluate the impact of genetic testing on healthcare decisions and patient outcomes in interventional pain management clinical care. Results of genetic testing will also be compared with the clinical outcome measures collected to discover novel genetic factors that may influence patient care.

DETAILED DESCRIPTION:
Specific genetic variations have been identified that result in alteration of expression or function of receptors, enzymes, and transporters that are relevant to the safety and efficacy of a medical treatment. By providing information regarding the genetic risks and the most effective therapy for an individual patient, clinicians may improve the efficacy of treatment and decrease the risk of adverse events.

The purpose of this study is to evaluate how currently available genetic tests are being implemented in various interventional pain management clinics around the United States, and whether this information results in benefits to patient care. Considering patient genotype correlates with pain sensitivity and perception, as well as autonomic nervous system dysfunction due to variations in sodium and potassium channels, genotypic associations can significantly improve outcomes in interventional pain management modalities including:

* Injections (also called nerve blocks using medications), such as steroids and opioids, including epidural steroid injections, facet joint injections, single nerve root blocks, and sacroiliac joint injections;
* Radiofrequency Rhizotomy (radiofrequency ablation and neuroablation), using x-ray guidance and a needle with an electrode at the tip that gets heated, to temporarily turn off a nerve's ability to send pain messages to the brain; and,
* Intrathecal pump implants which provide potent medications straight to the source of pain.

Patient that are receiving Proove Bioscience's genetic testing will complete validated questionnaires to measure specific outcomes related to their treatment at each clinical visit, including medication efficacy, reduction in adverse drug events, and healthcare utilization. Physicians will document any changes made to treatment regimens, including adjustments to medications or non-pharmacological treatments, and any improvements in the outcome measures. Statistical analysis will be performed to calculate relationships between genotypic and phenotypic data points collected in this study.

The results of this study will provide a measurable understanding of the medical and economic value of implementing genetic testing into interventional pain management. Furthermore, data points collected will be used to examine novel correlations and associations between single nucleotide polymorphisms and longitudinal clinical outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or Female, at least 18 years of age
* Currently taking or a candidate for opioid pain medication
* Documented or recent complaint of pain within 90 days (location to be documented in the case report form) with initial date of onset

Exclusion Criteria:

* Severe hepatic or renal disease (where current pharmaceutical dosing is affected and/or requires adjustment of standard dosing prior to PGx testing)
* Significant diminished mental capacity that is unable to understand the protocol, surveys and questionnaires; unable to read/write English or Spanish.
* Recent febrile illness that precludes or delays participation by more than 1 month
* Pregnancy or lactation
* Participation in a clinical study that may interfere with participation in this study
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be adult patients who are candidates for interventional pain management treatments, including Injections, Radio-frequency, Intrathecal pump implants, etc. All patients are receiving routine medical visits for their care and will have Proove laboratory genetic testing performed.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Pain Scores on the Pain Numeric Rating Scale (NRS) | 60 days
Function/Disability assessment on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 60 days
Number of Participants that Experience of Adverse Events | Up to 2 years
Type of Adverse Events Experienced by Participants | Up to 2 years
Severity of Adverse Events Experienced by Participants | Up to 2 years
Type of treatments selected for participants | 60 days
Medication dosage prescribed to the participants | 60 days
Frequency of participant urine drug screens | 60 days
Self-rated response levels to prescribed medications | 60 days

SECONDARY OUTCOMES:
Co-occurring disorders reported by ICD-9/10 code | 60 days
Assessment of previous treatments | 60 days
Urine drug screen results | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Maneesh Sharma, M.D., Principal Investigator — Interventional Pain Institute
Locations (31):
- United States (31):
  - Central Arizona Pain Institute, Prescott, Arizona
  - Spine Specialty Clinic of Arkansas, Heber Springs, Arkansas
  - Steven J. Waltrip M.D. Inc., Beverly Hills, California
  - Nuvo Spine, Encino, California
  - Memorial Orthopaedic Surgical Group, Long Beach, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Snibbe Orthopedics, Los Angeles, California
  - San Diego Pain Institute, San Diego, California
  - Dr. Anuj Gupta, Vista, California
  - Integrated Pain Solutions of South FL, Fort Lauderdale, Florida
  - Spinal Interventional Research, Gulf Breeze, Florida
  - Stuart B Krost MD, Lake Worth, Florida
  - Panama Interventional Pain Management, Panama City Beach, Florida
  - Interventional Pain Physicians of South Florida, Pembroke Pines, Florida
  - Neurological Spine & Pain, Savannah, Georgia
  - Wellspring Pain Solutions, Columbus, Indiana
  - Compass Pain Care, Charleston, South Carolina
  - Palmetto Pain Management, Columbia, South Carolina
  - Dr. Todd Joye, Mt. Pleasant, South Carolina
  - Coastal Interventional Pain Associates, Myrtle Beach, South Carolina
  - Pain, Spine and Sports Medicine, Myrtle Beach, South Carolina
  - Palmetto Spine and Pain Care Consultants, Myrtle Beach, South Carolina
  - El Paso Orthopaedic Surgery Group, El Paso, Texas
  - Medical Centre Pain Mgmt, Fort Worth, Texas
  - TX Spine and Joint, Houston, Texas
  - KSF Orthopaedic Center, Houston, Texas
  - North Hills Pain, Hurst, Texas
  - The Woodlands Pain Institute, Shenandoah, Texas
  - Victoria Pain and Rehabilitation Center, Victoria, Texas
  - National Spine And Pain Centers, McLean, Virginia
  - Northwest Spine and Pain Medicine, Spokane, Washington